CLINICAL TRIAL: NCT06695585
Title: Optimal Intravesical Lidocaine Volume for Pain Relief During Office Intra-detrusor Onabotulinum Toxin a Injections: a Prospective Randomized Superiority Trial
Brief Title: Optimal Intravesical Lidocaine Volume for Pain Relief During Office Intra-detrusor Onabotulinum Toxin a Injections
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Sean Francis, MD, OBGYN Department Chair, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 24.0636
Record Dates: First submitted 2024-11-11; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome; Urinary Urgency; Urinary Frequency; Urge Incontinence; Neurogenic Bladder
Keywords: Bladder Botox; Intravesical lidocaine; office Botox
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Bladder, Neurogenic | interventions — Lidocaine; onabotulinum toxin A

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded, randomized superiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Higher volume intravesical lidocaine (Active Comparator): 200 ml of 2% lidocaine without epinephrine intravesical instillation 20-30 minutes prior to bladder botox.
  Interventions: Drug: Lidocaine 2% without vessel constrictor
- Lower volume intravesical lidocaine (Active Comparator): 30 ml of 2% intravesical lidocaine without epinephrine instilled into the bladder 20-30 minutes prior to bladder botox.
  Interventions: Drug: Lidocaine 2% without vessel constrictor

INTERVENTIONS:
Drug: Lidocaine 2% without vessel constrictor — different volumes of intravesical 2% lidocaine without epinephrine, all patients will be receiving bladder botox but this will not be compared
  Other Names: onabotulinum toxin

SUMMARY:
The purpose of our study is to evaluate the efficacy and safety of different volumes of bladder-numbing medication for pain relief at the time of office bladder Botox injections. This is a randomized prospective, double-blind superiority trial comparing 200 ml 2% lidocaine versus 30 ml 2% lidocaine for office Botox injections.

DETAILED DESCRIPTION:
The volume of 2% intravesical lidocaine solution and efficacy for pain relief at the time of office intradetrusor Botox A injection has not been well studied. Studies evaluating intravesical lidocaine show that it is not sufficiently absorbed by human bladders to achieve serum toxicity levels and only provides superficial local anesthetic effect. Experts agree that intravesical local anesthetic can be given in the office, with approximately 30 to 40 mL of 2% lidocaine instilled via catheter into the bladder for about 20 minutes before injection. However, there is little evidence regarding this strategy, and future research would help standardize recommendations.

The purpose of our study is to evaluate the efficacy and safety of higher volume pre-procedure intravesical lidocaine solution for pain at the time of intradetrusor office Botox injections. This is a randomized prospective, double-blind superiority trial comparing 200 ml 2% lidocaine versus 30 ml 2% lidocaine for office Botox injections.

ELIGIBILITY:
Inclusion Criteria:

* Adult female, >18 years, English-speaking (surveys utilized are not validated in all languages)
* Able to provide informed consent
* Indications: Refractory urge urinary incontinence, Refractory urinary urgency and frequency, Neurogenic bladder (without sensory deficit)

Exclusion Criteria:

* Untreated urinary tract infection at the time of procedure
* Contra-indication to Botox
* Contraindication to intravesical lidocaine
* Inability to provide informed consent
* Pregnancy, breast-feeding, intending to become pregnant within 6 months of treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female anatomy
Enrollment: 36 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | on day of enrollment and procedure
  a. Determine the efficacy of pain relief via the Visual Analog Scale (VAS, scored 0-100 on 100 mm scale with 0 indicating no pain and 100 indicating the worst pain possible) in women randomized to 200 ml 2% lidocaine without epinephrine versus 30 ml 2% lidocaine without epinephrine prior to office intravesical onabotulinum toxin A (Botox) injections i. Perceived maximum VAS during the procedure and post-procedure ii. Superiority limit 20 mm on 100 mm VAS scale

SECONDARY OUTCOMES:
Patient Global Impression of Severity (PGI-S) | through study completion, an average of 1 year
  Likert scale describing current severity of urinary tract condition: 1. Normal, 2. Mild, 3. Moderate, 4. Severe; higher scores indicate worse symptoms
Overactive Bladder Satisfaction with Treatment Questionnaire (OAB-Sat-q) | This will be assessed pre and post-intervention for all participants through study completion, an average of 1 year
  An 11-item questionnaire that assesses patient satisfaction with their overactive bladder (OAB) treatment. It includes three sub-scales (satisfaction, side effects, and endorsement) and two single-item assessments (convenience and preference). Scores range from 0-100, higher scores indicate higher satisfaction with treatment. Used to assess treatment satisfaction over time.
Patient Satisfaction Questionnaire Short-Form (PSQ-18) | through study completion, an average of 1 year
  An 8-item question assessing satisfaction with medical care experience, measured on a Likert scale with 1 "Strongly agree" and 5 "Strongly disagree", for questions 1-3, 5-6, and 8 lower scores indicate higher satisfaction. For questions 4 and 7 lower scores indicate dissatisfaction.
Patient Global Impression of Improvement (PGI-I) | through study completion, an average of 1 year
  7-point Likert scale with 1 indicating "Very much better" and 7 indicating "Very much worse", lower scores indicate more improvement
Bladder diary | through study completion, an average of 1 year
  3-day bladder diary with objective patient reported data reporting voids per day, frequency between voids (measured in minutes or hours), episodes of incontinence per day
Post-void residual volume | through study completion, an average of 1 year
  Measure voided volume and obtain post-void residual volume either by bladder scan or straight catheterization in the office at 2-week follow up appointment (or additional time points if indicated) following bladder Botox injection
Adverse events | through study completion, an average of 1 year
  All adverse events will be recorded and tracked, including urinary tract infection, urinary retention, persistent hematuria, or additional suspected procedural related complications

CONTACTS AND LOCATIONS:
Overall Officials: Sean Francis, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Division of Urogynecology and Reconstructive Pelvic Surgery, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share data with other researchers/outside affiliates

REFERENCES:
- [Background] Nambiar AK, Younis A, Khan ZA, Hildrup I, Emery SJ, Lucas MG. Alkalinized lidocaine versus lidocaine gel as local anesthesia prior to intra-vesical botulinum toxin (BoNTA) injections: A prospective, single center, randomized, double-blind, parallel group trial of efficacy and morbidity. Neurourol Urodyn. 2016 Apr;35(4):522-7. doi: 10.1002/nau.22750. Epub 2015 Mar 8. PMID 25754188